CLINICAL TRIAL: NCT04306419
Title: Observational Trial on Cytokine Adsorption in Sepsis
Acronym: OuTCASt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Alexander Kersten, Principal Investigator, RWTH Aachen University
Other Study IDs: 19-058
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Sepsis; Septic Shock; Multiple Organ Failure
Keywords: Septic shock; cytokine adsorption therapy; HA-380 cartridge; Sepsis; hemoperfusion; multiple organ failure
MeSH Terms: conditions — Sepsis; Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the specific population of critically ill septic patients who benefit most from cytokine adsorption therapy with the HA-380 cartridge. Benefit of the treatment will be assessed on the basis of:

* The scope of the effect of cytokine adsorption therapy in this specific population of critically ill patients expressed by cytokine variability within the patients
* The scope of cytokine changes in passing the adsorption cartridge my measuring cytokine levels in the patient's blood directly before passing through the cartridge and directly after having passed through the cartridge.
* The scope of changes in organ dysfunction expressed by SOFA scores that are repeatedly calculated during the treatment with cytokine adsorption and then daily until day 7 of the ICU treatment.
* The scope of changes on cellular function on immune cells in serum samples taken before and after cytokine adsorption therapy.
* The scope of removal of anti-infective drugs from the blood in passing through the cytokine adsorption cartridge by measuring antibiotic drug levels in the patients blood during the cytokine adsorption therapy
* 30 day and 90 day mortality and location status in survivors

DETAILED DESCRIPTION:
1. Medical Problem Sepsis, a syndrome of physiologic, pathologic, and biochemical abnormalities induced by infection. It is a major public health concern, accounting for more than $20 billion (5.2%) of total US hospital costs in 2011. Sepsis has shown an increase in incidence most likely due to a combination of aging patient populations with more comorbidities and greater recognition. Sepsis is by conservative estimates a leading cause of mortality and morbidity in critical illness with long term sequelae for survivors.

   Underlying to sepsis is a multifaceted host response to an infecting pathogen that may be significantly amplified by endogenous factors and is defined by a nonhomeostatic, dysregulated host response to the infection with a potential lethality that is considerably in excess of that straightforward infection. In the early phases, an overshoot of pro-inflammatory mediators is often observed, caused by pathogen-associated molecular patterns (PAMPs) and damage-associated molecular patterns (DAMPs). High levels of pro- and anti-inflammatory cytokines are both associated with increased mortality. Blocking of overproduction of these cytokines using monoclonal anti- bodies targeting specific cytokines such as tumor necrosis factor-α (anti-TNF-α) have not demonstrated mortality benefits in larger trials.

   Therefore, an approach to decrease cytokine overproduction by using extracorporeal blood purification has previously been examined. Initial trials using Polymyxin B showed favorable results for markers of critical care treatment with a reduction of vasopressor dosage and higher ratios oxygen partial pressure to inspired oxygen. A larger randomized trial by Payenne however did not show any improvement of organ dysfunction or reduction in mortality by using Polymycin B hemoperfusion.

   A recent trial on the effect of the CytoSorb adsorption device using Interleucin-6 (IL-6) levels as marker of efficacy did also not find an effect of mortality, improved organ dysfunction or in fact a reduction of circulating IL-6 levels. However, in this trial the baseline cytokine levels were only moderately increased to begin with suggesting use of a device within a suboptimal patient population.

   As no more approved specific therapies to treat sepsis, exist following the withdrawal of recombinant activated protein C (Xigris; Eli Lilly, USA) from the market in 2011 following the results of the PROWESS-SHOCK trial and the pathophysiologic basis for mechanisms in sepsis due to an excess cytokine release are sound, the extracorporeal removal of cytokines remains a promising therapeutic target given the correct patient population.
2. Principal research question and novel aspects Within the trials addressing removal of excess cytokines, the selection of patients and timing of the intervention has been difficult, and results have not been conclusive. Data on the patient population which might benefit most in regard to the aspects of cytokine levels removed and organ failure or progressive organ dysfunction averted are sparse or non-existent. Even the largest randomised trial so far was active for 3 years in recruiting 100 patients out of 580 patients screened. This trial failed to show a positive effect on the primary endpoint of IL-6 removal as well as on secondary endpoints of morbidity or 30 day mortality. However, in this small trial there was a very low median cytokine level measured at baseline and randomisation which might be associated with the consecutive failure to detect a reduction in circulating cytokines. The question remains, whether this trial identified a patient population that was going to benefit from such a therapy to begin with. Post-hoc analyses of another trial, the Euphrates trial showed that there might be positive signal for reduced mortality in patients with an endotoxin activity that was in a mid-range and not at the highest end of the spectrum.

   We therefore aim to undertake an observational trial to examine the effect of treating sepsis according to the surviving sepsis campaign guidelines and using extracorporeal cytokine removal looking at circulating cytokine levels and development of new or worsening organ dysfunction in patients with sepsis or septic shock who show highly increased IL-6 levels.
3. HA 330 and HA 380 Hemoperfusion Cartridge The HA type resin cartridge (Jafron Industries, China) is an extracorporeal hemoperfusion device that uses neutral microporous resin, and it has been proven to specifically absorb different media- tors such as bilirubin and cytokines.

The HA380 HA 330 and HA 380 resin cartridges haves the ability to absorb various medium-sized factors, including most inflammatory cytokines (IL-1, IL-6, IL-8, IL-10 and TNF-a) and haves therefore lately been used in the treatment of patients with sepsis in China with several case reports demonstrating promising results on the clinical course of treated patients. Furthermore, there pooled there is emerging data that this therapeutic concept is efficienct and helpful in adequately selected patient populations.

The HA 380 cartridge is the CE-labeled updated version of the HA-330 cartridge which features a larger surface area of the resin beads increasing the overall capacity and thus potential efficacy of the device.

The HA 380 Hemoperfusion Cartridge works using Van der Waals interaction between resin molecular groups and adsorbed substances. Unlike the CytoSorb device, these are incorporated into the resin molecule by a molecular sieve effect of the 3D network structure and the lipophilic hydrophobicity of the molecular group. Therefore, the pass-through effect in removing cytokines is expected to be larger and more sustained, as previously adsorbed cytokines will not again be released by continued blood flow or movement of the device. The range of adsorption is shown in figure 1. The device described has a CE label and is approved for treatment in a variety of clinically situations including but not limited to intra-operative use in cardiac surgery, intoxication, liver failure and sepsis. Compared to other available devices which could be used in the same settings this cartridge offers superior flow characteristics, less flow resistance and a higher capacity of cytokine removal. The effect of combining a standard treatment course of sepsis according to the Surviving Sepsis Campaign guidelines with extracorporeal cytokine removal however is not well examined overall.

In the investigator center, the investigators have therefore undertaken a retrospective pilot observational trial of 15 patients in which the using the HA 380 330 device was used as a rescue therapy in therapy in 15 patients with septic shock and multi-organ failure refractory to conventional treatment. In this trial of extremely ill patients the investigators found a significant difference between hospital survivors and non-survivors in circulating IL-6, IL-10 and TNF-alpha levels after 8 hours of treatment with the HLA 3380 cartridge. However, the overall variation of cytokine levels at baseline and the variation of changes from baseline during therapy were rather large. The sample size was too small to infer any causality or undertake multi-variate analysis.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. diagnosis of sepsis or septic shock with at least 2 organ-dysfunctions defined by SOFA score
3. baseline serum IL-6 > 1000 pg/ml, IL-10 levels >250 pg/ml or TNF-alpha levels > 100 ng/l. The baseline IL-6 measurement must be on the same calendar day that the cytokine adsorption is started, the baseline IL-10 or TNF-alpha can be taken up to 36h before because of higher turn-around times for these tests.
4. need for CRRT or ECMO therapy

Exclusion Criteria:

1. Solid organ malignancies with or without treatment
2. Participation or enrollment in another clinical study within 30 day
3. Pregnant and lactating females If women of childbearing potential will be enrolled, a pregnancy test will be performed by assessing the value of ß-HCG in the routinely drawn blood and or urine.
4. Patient has been committed to an institution by legal or regulatory order
5. Participation in a parallel interventional clinical trial
6. The subject received an investigational drug within 30 days prior to inclusion into this project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will perform an observational trial in a large cohort of patients with sepsis and septic shock who are treated with cytokine adsorption by hemoperfusion with a HA-380 cartridge. Sepsis will be defined as done in the Sepsis-3 definition. In addition to sepsis or septic shock patients must have a confirmed excess of IL-6, IL-10 or TNF-alpha or a combination of these with IL-6 levels > 1000 pg/l, IL-10 levels >250 pg/l or TNF-alpha levels > 100 ng/l. Patients must be in need of CRRT or ECMO therapy to perform the HA-380 therapy. Stand-alone hemoperfusion will not be performed.
  Patients must be included within 24 hrs of diagnosing sepsis. The IL-6 measurement for inclusion must be from within 24 hrs, IL-10 or TNF-alpha measurements for inclusion can be from within 36 hrs before inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-06-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Cytokine variability of Interleucin (IL) -6 , IL-8- IL-10, and Tumor Necrosis Factor-alpha (TNF-alpha) in the patient's IL-6 serum | 16 hours
  as expressed by changes in concentration measured every two hours during a first cytokine adsorption treatment of eight hours and measured every four hours during a second eight hour cytokine adsorption treatment. The measurements will be set in relation to the baseline measurement taken immediately (<1 minute) immediately after the end of 8 hours of treatment with the HA 380 cartridge normalized to the initial baseline IL-6 serum concentration immediately before start of the treatment. The standard of care is a pause of four hours between the two treatments intervals

SECONDARY OUTCOMES:
Efficacy of relative cytokine removal from the patient's blood | 20 hours
  by measuring relative differences for IL-6 , IL-8- IL-10 and TNF-alpha in blood samples taken directly before the blood enters the cartridge (inflow) and directly after passing the cartridge (outflow) during the treatments with the HA-380 cartrdige at the timepoints T2, T4, T6, T8 and T12, T16, T20.
Vasopressor / lactate dose | 8 hours
  Normalized change in vasopressor dose and lactate from baseline to after each 8 hours of treatment with the HA 380 cartridge
P/F ratio | 8 hours
  Normalized change in P/F ratio from baseline to after each 8 hours of treatment with the HA 380 cartridge
Antibiotic drug levels | 20 hours
  Changes in antibiotic drug levels between T0, T8 and T20 taken from the patient's blood samples at these time points.
Sequential Organ Failure Assessment (SOFA) | 3 hours
  Individual SOFA score changes and total SOFA Score changes over the course of each 8 hour treatment and the interval between the two treatments (T0,T2,T4,T6,T8,T12,T16,T20), and afterwards daily for a maximum of 7 days after the HA-380 treatment, until death of the patient or t until the patient leaves the ICU for, whichever occurs first.
  breathing activity (minimum <100 mmHg gets 4 Points; maximum <400 gets 1 Points; higher Points means a worse outcome)
  Liver function (minimum 1,2 mg/dl of Bilirubin gets 1 Points; maximum >12 mg/dl Bilirubin gets 4 Points; higher Points means a worse outcome)
  Blood Coagulation (minimum <20 Thrombocyten x10^3/µl gets 4 Points; maximum >150 Thrombocyten x10^3/µl gets 4 Points; higher Points means a worse outcome)
  Renal function (minimum 1,2 mg/dl of Kreatinin gets 1 Points; maximum >5 mg/dl Kreatinin gets 4 Points; higher Points means a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Torio CM, Andrews RM. National Inpatient Hospital Costs: The Most Expensive Conditions by Payer, 2011. 2013 Aug. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #160. Available from http://www.ncbi.nlm.nih.gov/books/NBK169005/ PMID 24199255
- [Background] Gaieski DF, Edwards JM, Kallan MJ, Carr BG. Benchmarking the incidence and mortality of severe sepsis in the United States. Crit Care Med. 2013 May;41(5):1167-74. doi: 10.1097/CCM.0b013e31827c09f8. PMID 23442987
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Vincent JL, Marshall JC, Namendys-Silva SA, Francois B, Martin-Loeches I, Lipman J, Reinhart K, Antonelli M, Pickkers P, Njimi H, Jimenez E, Sakr Y; ICON investigators. Assessment of the worldwide burden of critical illness: the intensive care over nations (ICON) audit. Lancet Respir Med. 2014 May;2(5):380-6. doi: 10.1016/S2213-2600(14)70061-X. Epub 2014 Apr 14. PMID 24740011
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Kellum JA, Kong L, Fink MP, Weissfeld LA, Yealy DM, Pinsky MR, Fine J, Krichevsky A, Delude RL, Angus DC; GenIMS Investigators. Understanding the inflammatory cytokine response in pneumonia and sepsis: results of the Genetic and Inflammatory Markers of Sepsis (GenIMS) Study. Arch Intern Med. 2007 Aug 13-27;167(15):1655-63. doi: 10.1001/archinte.167.15.1655. PMID 17698689
- [Background] Abraham E, Wunderink R, Silverman H, Perl TM, Nasraway S, Levy H, Bone R, Wenzel RP, Balk R, Allred R, et al. Efficacy and safety of monoclonal antibody to human tumor necrosis factor alpha in patients with sepsis syndrome. A randomized, controlled, double-blind, multicenter clinical trial. TNF-alpha MAb Sepsis Study Group. JAMA. 1995 Mar 22-29;273(12):934-41. PMID 7884952
- [Background] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Background] Payen DM, Guilhot J, Launey Y, Lukaszewicz AC, Kaaki M, Veber B, Pottecher J, Joannes-Boyau O, Martin-Lefevre L, Jabaudon M, Mimoz O, Coudroy R, Ferrandiere M, Kipnis E, Vela C, Chevallier S, Mallat J, Robert R; ABDOMIX Group. Early use of polymyxin B hemoperfusion in patients with septic shock due to peritonitis: a multicenter randomized control trial. Intensive Care Med. 2015 Jun;41(6):975-84. doi: 10.1007/s00134-015-3751-z. Epub 2015 Apr 11. PMID 25862039
- [Background] Schadler D, Pausch C, Heise D, Meier-Hellmann A, Brederlau J, Weiler N, Marx G, Putensen C, Spies C, Jorres A, Quintel M, Engel C, Kellum JA, Kuhlmann MK. The effect of a novel extracorporeal cytokine hemoadsorption device on IL-6 elimination in septic patients: A randomized controlled trial. PLoS One. 2017 Oct 30;12(10):e0187015. doi: 10.1371/journal.pone.0187015. eCollection 2017. PMID 29084247
- [Background] Ranieri VM, Thompson BT, Barie PS, Dhainaut JF, Douglas IS, Finfer S, Gardlund B, Marshall JC, Rhodes A, Artigas A, Payen D, Tenhunen J, Al-Khalidi HR, Thompson V, Janes J, Macias WL, Vangerow B, Williams MD; PROWESS-SHOCK Study Group. Drotrecogin alfa (activated) in adults with septic shock. N Engl J Med. 2012 May 31;366(22):2055-64. doi: 10.1056/NEJMoa1202290. Epub 2012 May 22. PMID 22616830
- [Background] Dellinger RP, Bagshaw SM, Antonelli M, Foster DM, Klein DJ, Marshall JC, Palevsky PM, Weisberg LS, Schorr CA, Trzeciak S, Walker PM; EUPHRATES Trial Investigators. Effect of Targeted Polymyxin B Hemoperfusion on 28-Day Mortality in Patients With Septic Shock and Elevated Endotoxin Level: The EUPHRATES Randomized Clinical Trial. JAMA. 2018 Oct 9;320(14):1455-1463. doi: 10.1001/jama.2018.14618. PMID 30304428
- [Background] Hu XB, Gao HB, Liao ME, He MR. [The use of HA330-II microporous resin plasma adsorption in the treatment of chronic severe hepatitis]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2007 Dec;19(12):760-1. No abstract available. Chinese. PMID 18093442
- [Background] Li G, Yang B, Li C, Chen Y, Guo X, He B, Zhang Y, Dai R. [Studies on adsorption of the organic phosphorus pesticide with the macroporous resin]. Sheng Wu Yi Xue Gong Cheng Xue Za Zhi. 2000 Dec;17(4):369-72. Chinese. PMID 11211815
- [Background] Gruda MC, Ruggeberg KG, O'Sullivan P, Guliashvili T, Scheirer AR, Golobish TD, Capponi VJ, Chan PP. Broad adsorption of sepsis-related PAMP and DAMP molecules, mycotoxins, and cytokines from whole blood using CytoSorb(R) sorbent porous polymer beads. PLoS One. 2018 Jan 25;13(1):e0191676. doi: 10.1371/journal.pone.0191676. eCollection 2018. PMID 29370247
- [Background] Bonavia A, Groff A, Karamchandani K, Singbartl K. Clinical Utility of Extracorporeal Cytokine Hemoadsorption Therapy: A Literature Review. Blood Purif. 2018;46(4):337-349. doi: 10.1159/000492379. Epub 2018 Sep 3. PMID 30176653